CLINICAL TRIAL: NCT05538988
Title: An Interventional, Single-arm, Open-label Phase I/II Study Investigating the Efficacy and Safety of Anti-PD1 Immunotherapy for the Treatment of Patients With Cutaneous T-cell Lymphoma (Mycosis Fungoides)
Brief Title: BIOmarker-guided Study to Evaluate the Efficacy and Safety of cemipLimab for advancEd Cutaneous T-cell Lymphoma
Acronym: BIOSELECT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Contractual Issues
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0028
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cemiplimab (Experimental): Study treatment includes administration of cemiplimab 350 mg intravenous every 21 days (+/﹣ 3 days)
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab is a recombinant human IgG monoclonal antibody known as a programmed cell death 1 (PD-1) immune checkpoint inhibitor. The PD-1 pathway is an immune system checkpoint that may be exploited by tumour cells to escape active T-cell surveillance. Cemiplimab binds to PD-1 on T cells and blocks the interaction with its ligands, PD-L1 and PD-L2. Inhibition of the receptor/ligand signaling restores the anti-tumour immune response
  Other Names: Libtayo

SUMMARY:
Background - Advanced cutaneous T-cell lymphoma (mycosis fungoides, MF) is an incurable extranodal mature lymphoma with poor prognosis. Currently available therapies provide only short-term remissions.

Rationale - MF is an immunogenic cancer and expresses a high number of neoantigens. therefore it it reasonable to assume that it would respond to immune checkpoint inhibitors.

Objectives - The primary objective is to test the clinical efficacy (objective response rate) of the immune checkpoint inhibitor cemiplimab in patients with advanced mycosis fungoides (MF) who failed first-line therapy, defined as the sum of complete and partial responses (where at least 50% reduction of mSWAT is achieved).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmation of mycosis fungoides; diagnosis must be confirmed by the Northern Alberta Cutaneous Lymphoma Review Board.
2. Minimum disease stage(s) for enrolment: stage IIB (see appendix B).
3. Patients must be 18 years of age or older.
4. Patients must be capable of providing consent to enrolment and willing to comply with study treatment and follow-up.
5. Patients with a performance status of ECOG 0-2(11) will be eligible for enrolment (see appendix A).
6. Previous failure of ≥1 prior therapies, including PUVA (psoralen and UVA phototherapy), systemic interferon α, systemic retinoid therapy (bexarotene, alliretinoin or acitretin), systemic histone deacetylase (HDAC) inhibitor (vorinostat or romidepsin), radiation therapy or systemic chemotherapy (including, but not limited to methotrexate and gemcitabine).
7. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
8. Patients of childbearing/reproductive potential should use adequate birth control methods, as defined by the investigator, during the study treatment period and for a period of 30 days after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
9. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
10. The following adequate organ function laboratory values must be met:

    a. Hematological: i. Absolute neutrophil count (ANC) ≥ 1,500 /mcL ii. Platelet count ≥100,000 / mcL iii. Hemoglobin >90 mg/dL (transfusions are permitted) b. Renal serum creatinine or (measured or calculated) creatinine clearance (GFR can also be used in place of creatinine or CrCl)≤1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels >1.5 X institutional ULN c. Hepatic: i. Total serum bilirubin <1.5 x ULN ii. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN

Exclusion Criteria:

1. Known immunodeficiency (including known history of human immunodeficiency virus (HIV)).
2. Active Hepatitis B or Hepatitis C. Testing for HBV or HCV is not mandatory for enrolment to study, but may occur at the discretion of the investigator. Inactive HBsAg carriers with prophylactic antiviral agent are allowed.
3. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids doses >20 mg daily for more that 2 months, or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Patients who have been previously treated with a PD(L)-1 immune checkpoint inhibitor regimen are ineligible.
5. Patients with a requirement for concomitant radiation therapy are ineligible; prior treatment with radiation therapy is not exclusionary, but a wash-out period of no less than 28 days is required prior to study enrolment.
6. Patients receiving immunosuppressive agents within 30 days prior to the first dose of trial treatment, including non-steroid immunosuppressive agents (e.g. anti-TNFα biologic agents, methotrexate, mycophenolate mofetil, tacrolimus) or systemic corticosteroids.
7. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class II) or serious cardiac arrhythmia requiring medication.
8. Presence of a concurrent (synchronous) second primary malignancy.
9. Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on the investigator's judgment are acceptable.
10. Known prior severe hypersensitivity to study drugs or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | The analysis of the primary endpoint will occur 90 days after 16 patients complete week 27 assessments.
  Efficacy of treatment will be described by an objective response rate (ORR) >50%. I.e. achieving ORR in 50% of the patients.

SECONDARY OUTCOMES:
Assessment of Treatment Safety | Adverse events will be reviewed throughout the study and the analysis will be completed 90 days following the 99 week follow-up.
  CTCAE v5.0 will be used to categorize treatment related and non-treatment related adverse events.
Assessment of Progression Free Survival (PFS) | The PFS analysis will be completed 90 days following the 99 week follow-up.
  Progression-free survival is defined as the time between the date of treatment initiation and the date of disease progression or death
Reduction in mSWAT during Therapy. | mSWAT will be assessed during screening, week 12, week 27, week 39 and week 48
  Clinical investigator will assess the patches, plaques and tumors on your skin and assign a value using a grid point system. These values will be assessed in relation to the original baseline value.
Duration of Objective Response to Therapy | The duration of objective response to therapy analysis will be completed 90 days following the 99 week follow-up.
  Duration of treatment response is defined as the elapsed time between demonstration of an objective response and subsequent progression of disease or censoring.
Health Related Quality of Life (EuroQol-5D) | The EuroQol-5D questionnaire will be administered at screening, Cycle 1 (each cycle is 21 days) and every 12 weeks (cycle 5, 9, etc. )thereafter until end of treatment (max of 17 cycles)
  The patient is asked to indicate his/her health state by ticking a box next to a series of questions. This decision results in a number that can be combined with the other questions to form a number that describes the patient's health state.
Health Related Quality of Life (Brief Older People's Quality of Life) | The OPQOL-Brief questionnaire will be administered at screening, Cycle 1 (each cycle is 21 days) and every 12 weeks (cycle 5, 9, etc. )thereafter until end of treatment (max of 17 cycles)
  The patient is asked to indicate his/her health state by ticking a box next to a series of questions. This decision results in a number that can be combined with the other questions to form a number that describes the patient's health state.
Health Related Quality of Life (Dermatological Life Quality Index) | The DLQI questionnaire will be administered at screening, Cycle 1 (each cycle is 21 days) and every 12 weeks (cycle 5, 9, etc. )thereafter until end of treatment (max of 17 cycles)
  The patient is asked to describe their skin problems by ticking a box next to a series of questions. This decision results in a number that can be combined with the other questions to form a number that describes how the patients skin problems have affected their quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided